CLINICAL TRIAL: NCT07405385
Title: Cardiotoxicity Assessment and Reduction Through Exercise in BREAST Cancer
Acronym: CARE-BREAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Susana Aznar Laín, Full professor, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-UNIVERS-12844
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Breast Cancer; Neoplasm; Cardiotoxicity
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Cardiotoxicity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE GROUP (Experimental)
  Interventions: Behavioral: Exercise
- CONTROL GROUP (Other)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Participants assigned to the control group receive standard care typically provided to patients in this phase of recovery. Instead of a supervised exercise program, these individuals are sent educational materials via email. This material consists of a video and official documents containing basic guidelines and recommendations for a healthy lifestyle, based on standards from the World Health Organization (WHO) and the American College of Sports Medicine (ACSM) for cancer survivors. The documents provide general instructions on physical activity, reducing sedentary behavior, and maintaining overall health habits. Like the intervention group, participants in the control group undergo all clinical and functional evaluations at the start of the study, after 16 weeks, and during a 3-month follow-up.
  Arms: CONTROL GROUP
Behavioral: Exercise — The intervention consists of a supervised, in-person, combined exercise program lasting 16 consecutive weeks, conducted at a specialized exercise unit. Participants attend two sessions per week, with at least 48 hours of recovery between sessions, and each session lasts between 55 and 85 minutes. The program follows a "combined" methodology, meaning every session integrates both resistance (strength) and aerobic training. To ensure safety and precision, sessions are led by a graduate in Physical Activity and Sport Sciences with specialized training in oncology, and participants work in small groups of 6 to 8 people.
  Each session is structured into four distinct parts: a 10-minute warm-up involving low-to-moderate intensity activity and joint mobility; a resistance training block; an aerobic training block; and a cool-down featuring static stretching for 30-40 seconds per muscle group. The resistance training portion utilizes a "full body" approach.
  Arms: EXERCISE GROUP

SUMMARY:
The CARE-BREAST study is a randomized, controlled clinical trial designed to evaluate the cardioprotective effects of a supervised exercise program in breast cancer survivors. Many life-saving breast cancer treatments, such as anthracyclines and targeted therapies like trastuzumab, are known to be cardiotoxic, potentially causing long-term damage to the heart and a significant decline in cardiorrespirator fitness. This damage, known as Cancer Therapy-Related Cardiac Dysfunction (CTRCD), can manifest months or even years after treatment ends, with the highest risk occurring during the first year of survivorship. This trial focuses on a critical "recovery window," recruiting women aged 30 to 70 who completed cardiotoxic treatments between six months and one year prior to joining the study.

The study operates on the primary hypothesis that breast cancer survivors who complete a 16-week supervised, combined exercise program will show significant improvements in myocardial function-specifically measured through the Left Ventricular Ejection Fraction (LVEF) and Global Longitudinal Strain (GLS)-as well as overall aerobic capacity (VO2max) when compared to a control group. The trial aims to determine if structured exercise can mitigate the subclinical heart damage caused by chemotherapy and improve the patient's physical health and quality of life during the transition to long-term survivorship.

Participants are randomly assigned to one of two groups. The intervention group participates in a 16-week program consisting of two weekly supervised sessions at a specialized exercise unit. Each session, lasting between 55 and 85 minutes, includes a combination of strength training and aerobic exercise tailored to each participant's individual fitness level. The control group receives standard educational materials via email regarding healthy lifestyle habits and exercise guidelines for cancer survivors but does not participate in the supervised training sessions.

To measure the study's impact, all participants undergo comprehensive medical evaluations before and after the 16-week period, including heart imaging via echocardiogram, blood tests to check for cardiac biomarkers like troponin, and a maximal exercise test to assess lung and heart capacity. By comparing these results between the two groups, the research team hopes to generate high-quality evidence that can be used to establish specific exercise prescriptions as a standard part of follow-up care for breast cancer survivors, ultimately helping to protect their heart health and improve their long-term survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 70 years.
* Confirmed diagnosis of breast cancer in stages I to III.
* Patients who completed treatment with cardiotoxic agents (anthracyclines, trastuzumab, or pertuzumab) between 6 months and 1 year prior to enrollment.
* Residency within a distance of less than 40 km from the Hospital Universitario de Toledo.

Exclusion Criteria:

* Diagnosis of diabetes mellitus with poor glycemic control, defined as an HbA1c value greater than or equal to 8.5%.
* Presence of an acute infectious disease.
* Medical contraindication for the performance of a maximal exercise stress test.
* Medical contraindication for the practice of physical exercise.
* Relative or absolute contraindications for physical exercise according to ACSM (American College of Sports Medicine) guidelines.
* Serious heart or cardiovascular disease, including a history of myocardial infarction, heart failure, or known cardiomyopathy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Global Longitudinal Strain | 7 months
  Measurement of myocardial deformation using transthoracic echocardiography to detect subclinical alterations in cardiac function.
Change in LVEF | 7 months
  Assessment of the volume of blood pumped out of the left ventricle with each contraction, measured via the biplane Simpson's method and 3D echocardiography.
Changes in Cardiorespiratory Fitness | 7 months
  Assessment of cardiorespiratory capacity determined through a maximal cardiopulmonary exercise test (stress test) on a cycle ergometer

SECONDARY OUTCOMES:
Change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) | 7 months
  Analysis of NT-proBNP levels via blood samples to evaluate cardiac wall stress.
Change in High-sensitivity Cardiac Troponin (hs-cTn) | 7 months
  Analysis of high-sensitivity cardiac troponin levels via blood samples to identify myocardial injury.
Change in Lower Body Muscular Strength | 7 months
  Estimated one-repetition maximum (1RM) for the leg press. Measurements will be obtained through force-velocity profiling using a linear position transducer.
Change in Upper-Body Muscular Strength | 7 months
  Estimated one-repetition maximum (1RM) for the vertical press. Measurements will be obtained through force-velocity profiling using a linear position transducer.
Change in 6-Minute Walk Test | 7 months
  Evaluation of physical performance using the 6-minute walk test.
Change in Lower-Body Muscular Endurance (30-sec CST) | 7 months
  Evaluation of physical performance using the 30-second chair stand test.
Change in Grip Strength | 7 months
  Evaluation of upper-body isometric strength using a handheld dynamometer.
Change in Body Mass Index (BMI) | 7 months
  BMI will be calculated as weight in kilograms divided by height in meters squared (kg/m2).
Change in Body Fat Percentage | 7 months
  Assessment of total body fat percentage using bioelectrical impedance analysis (BIA).
Change in Lean Mass Percentage | 7 months
  Assessment of total lean muscle mass percentage using bioelectrical impedance analysis (BIA).
Change in Bone Mass | 7 months
  Assessment of estimated bone mineral mass using bioelectrical impedance analysis (BIA).
Change in EQ-5D-5L Visual Analogue Scale (VAS) | 7 months
  Evaluation of self-rated health using the EuroQol Visual Analogue Scale (EQ VAS). The scale is a vertical line with minimum value 0 (worst imaginable health) and maximum value 100 (best imaginable health). Higher scores indicate a better perceived health outcome.
Change in EQ-5D-5L Index Score | 7 months
  Evaluation of health-related quality of life based on the EuroQol 5-dimension 5-level (EQ-5D-5L) descriptive system. This system assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses are converted into a single index score using a valuation algorithm. The index scale typically ranges from less than 0 to 1, where higher scores indicate a better outcome.
Change from Baseline in Cancer-Related Fatigue (FACIT-F) | 7 months
  Evaluation using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale. Total scores range from 0 to 52, where higher scores indicate lower levels of fatigue.
Change in Hospital Anxiety and Depression Scale (HADS) | 7 months
  Evaluation using the Hospital Anxiety and Depression Scale (HADS). The total score ranges from 0 to 42, where higher scores indicate greater psychological distress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Castilla-La Mancha (PAFS Research Group), Toledo, Toledo, Spain